CLINICAL TRIAL: NCT07406594
Title: MICRO-VERZ: MICRObiome Changes During VERZenio Therapy
Brief Title: Gut Microbiome Changes During Abemaciclib Therapy in Breast Cancer
Acronym: MICRO-VERZ
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vermont Medical Center (Other)
Responsible Party: Principal Investigator, Tracy Smith, Faculty Scientist, University of Vermont Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MICRO-VERZ
Record Dates: First submitted 2026-01-27; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Breast Cancer; HER-2 Positive Breast Cancer
Keywords: microbiome
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resistant Starch Intervention (Experimental): Participants randomized to this arm will receive resistant starch powder as a dietary supplement during early abemaciclib therapy. The supplement will be taken orally as a powder mixed with a beverage, according to instructions provided. Participants will continue to receive abemaciclib as standard of care and will complete study procedures including stool sample collection and symptom questionnaires.
  Interventions: Dietary Supplement: Resistant Potato Starch
- Placebo Supplementation (Control Arm) (Placebo Comparator): Participants randomized to this arm will receive a placebo powder as a dietary supplement during early abemaciclib therapy. The placebo will be taken orally as a powder mixed with a beverage, according to instructions provided. Participants will continue to receive abemaciclib as standard of care and will complete study procedures including stool sample collection and symptom questionnaires.
  Interventions: Dietary Supplement: Placebo control

INTERVENTIONS:
Dietary Supplement: Resistant Potato Starch — Participants randomized to the resistant starch intervention will receive a resistant starch dietary supplement administered orally. The supplement will be taken during early abemaciclib therapy according to study instructions. Abemaciclib is administered as standard of care and is not altered by study participation.
  Arms: Resistant Starch Intervention
Dietary Supplement: Placebo control — Participants randomized to the placebo intervention will receive a placebo dietary supplement administered orally as a powder mixed with a beverage. The supplement will be taken during early abemaciclib therapy according to study instructions. Abemaciclib is administered as standard of care and is not altered by study participation.
  Arms: Placebo Supplementation (Control Arm)

SUMMARY:
Abemaciclib (Verzenio) is a commonly used treatment for hormone receptor-positive breast cancer, but it can cause gastrointestinal side effects such as diarrhea, which may affect quality of life and treatment tolerance. The gut microbiome, which is the collection of bacteria living in the digestive tract, may play a role in these symptoms.

The purpose of this study is to examine how the gut microbiome changes during the early phase of abemaciclib treatment and how these changes relate to gastrointestinal symptoms experienced by patients. Participants will provide stool samples at multiple time points using mailed collection kits and will complete questionnaires about gastrointestinal symptoms while receiving standard-of-care abemaciclib therapy. All study procedures will be conducted remotely.

Information gained from this study may help inform future supportive care strategies for breast cancer patients receiving abemaciclib.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Histologically confirmed hormone receptor-positive, HER2-negative breast cancer.
* Planned initiation of adjuvant abemaciclib (Verzenio) as part of standard clinical care, with enrollment occurring prior to or within 7 days of starting abemaciclib.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
* Women of child-bearing potential must agree to use contraception prior to study entry, for the duration of study participation, and for 90 days following completion of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

A female of child-bearing potential is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

* Has not undergone a hysterectomy or bilateral oophorectomy; or
* Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months).

  * Ability to understand and the willingness to sign a written informed consent.

Exclusion Criteria:

* Concurrent participation in another interventional clinical trial that, in the opinion of the investigator, would interfere with study participation or interpretation of results.
* Known gastrointestinal conditions that would significantly interfere with study procedures or interpretation of results, including but not limited to inflammatory bowel disease, short bowel syndrome, or chronic diarrheal disorders.
* Known allergy or intolerance to resistant starch or any component of the study supplement.
* Pregnant or breastfeeding individuals.
* Any medical, psychiatric, or social condition that, in the judgment of the investigator, would limit the participant's ability to comply with study procedures.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2027-10 (Estimated); Primary Completion 2031-10 (Estimated); Study Completion 2031-10 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | From study opening through completion of enrollment (approximately 12 months)
  Feasibility will be assessed by the proportion of eligible participants who enroll in the study out of those approached for participation.
Participant retention | Through end of intervention (6 weeks)
  Feasibility and acceptability will be assessed by the proportion of enrolled participants who complete the intervention period and final study assessments.
Supplement adherence | During the 6-week intervention
  Feasibility will be assessed by participant adherence to the assigned supplement, measured as the proportion of prescribed doses taken during the intervention period.
Completion of study procedures | Baseline through end of intervention (6 weeks)
  Feasibility will be assessed by the proportion of participants who complete protocol-specified stool sample collections and questionnaires.

SECONDARY OUTCOMES:
Change in Gut Microbial Community Composition During Early Abemaciclib Therapy | Baseline through Week 6 of abemaciclib therapy
  Changes in gut microbial community composition will be assessed using stool samples collected at baseline and during early abemaciclib therapy. Microbiome profiles will be compared over time and between intervention groups to characterize longitudinal changes associated with treatment.
Correlation between gut microbiome diversity and gastrointestinal symptom severity | Baseline through Week 6 of abemaciclib therapy
  Correlation between gut microbiome alpha diversity measured from stool samples using 16S rRNA gene sequencing (Shannon diversity index, unitless) and gastrointestinal symptom severity measured using the Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE) gastrointestinal symptom items (score range 0-4 per item). Correlation coefficients will be calculated to assess the relationship between microbiome diversity and symptom severity during early abemaciclib therapy.
Differences in Gut Microbial Community Composition Between Resistant Starch and Placebo Groups | Baseline through Week 6 of abemaciclib therapy
  Differences in gut microbial community composition and temporal patterns will be explored between participants randomized to resistant starch supplementation and those receiving placebo using stool samples collected at multiple time points during early abemaciclib therapy.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Vermont, Burlington, Vermont, United States

IPD SHARING:
Plan to Share IPD: Undecided